CLINICAL TRIAL: NCT05718661
Title: The Effectiveness of Virtual Reality Distraction on Preoperative Anxiety in Abdominal Surgery Patients: A Double-Blinded Randomised Controlled Trial
Brief Title: The Effect of Virtual Reality Distraction on Preoperative Anxiety in Abdominal Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sevim Akbal, Assistant Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TUTF-GOBAEK 2022/240
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Anxiety
Keywords: virtual reality; abdominal surgery; randomised controlled trial
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This research was designed using the experimental (intervention) research method. Under the same environment and conditions, to determine the effect on the same dependent variable, the intervention (experimental) group using virtual reality and the placebo group not using virtual reality (watching the same video with the naked eye), pre-test (measurement of the dependent variable before the intervention), post-test (dependent measurement of the variable after intervention). In addition, the group that was not interfered with will form the control group and a data collection form will be applied with an interval of 30 minutes.
Who Masked: Participant, Investigator
Masking Description: The evaluation process consisted of two stages: the first evaluation conducted in the morning and the second evaluation performed immediately before the patients were transferred to the operating room. To maintain blinding during the data collection, the patient information, anxiety and stress levels of the patients were evaluated by three senior nursing student researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses Group (Experimental): The intervention group will watch a virtual reality video with mobile virtual glasses by the researcher (SŞ) and the stress level on the smart wristband will be recorded. In addition, necessary variables will be recorded with the data collection form.
  Interventions: Behavioral: Watching video with virtual glasses
- Non-Virtual Reality Glasses Group (Placebo Comparator): The plain version of the video, which was shown to the intervention group by the researcher (SŞ) to the placebo group, will be watched over the phone with the naked eye and the stress level on the smart bracelet will be recorded. In addition, necessary variables will be recorded with the data collection form.
  Interventions: Behavioral: watching video without virtual glasses
- Control Group (No Intervention): Anxiety control will be done by the researcher (SU) for the control group.

INTERVENTIONS:
Behavioral: Watching video with virtual glasses — Using Mobile Virtual Glasses; In the preoperative period, after the patient is taken to the surgical service, a virtual reality video will be watched with mobile virtual glasses at the specified time (before going to the operating room on the day of surgery). Measurements will be made before and after the application. Necessary hygiene will be provided before the use of glasses, and the researcher will ensure hand cleaning before entering the patient's room.
  Arms: Virtual Reality Glasses Group
Behavioral: watching video without virtual glasses — The plain version of the video, which was shown to the intervention group by the researcher (SŞ) to the placebo group, will be watched over the phone with the naked eye and the stress level on the smart bracelet will be recorded.
  Arms: Non-Virtual Reality Glasses Group

SUMMARY:
Hospitalization, medical interventions to be performed, and uncertainties specific to surgical intervention create a certain level of anxiety in the patient. It is known that being in the hospital negatively affects the coping mechanisms of the patient. In the pre-surgical period, the nurse's practices that will facilitate the patient's coping with the situation and managing his anxiety have a positive effect on anxiety during and after surgery and on anxiety-related symptoms. For these reasons, it is aimed to determine the effect of virtual reality on pre-surgical anxiety in this study.The hypothesis of the study is that watching videos with virtual glasses will reduce preoperative anxiety.

DETAILED DESCRIPTION:
Hypothesis H1: The anxiety level of patients who watch relaxing video through VR is lower than that of those who do not.

H2: The stress level of patients who watch relaxing video through VR is lower than that of those who do not.

H3: The heart rate level of patients who watch relaxing video through VR is lower than that of those who do not.

This study was carried out between January 30, 2023 and December 20th 2024 at the General Surgery Service of a university hospital, which has a 48-bed capacity and accommodates 1-2 patients per room. The hospital is situated in the Trakya region of the Edirne province in Türkiye and serves as a major healthcare provider, offering a comprehensive range of medical services to the surrounding provinces and contributes to medical and health sciences education and research. At this service, nurses ensure that patients are prepared for surgery in accordance with the daily determined operating room schedule by instructing them to remove their clothing, except for their underwear, and put on their green surgical gowns and caps. Following this preparation, patients remain in their beds while awaiting the arrival of healthcare support personnel for their transfer to the operating room. This waiting period typically lasts between 20 to 25 minutes.

The sample size was calculated based on the study by Mosso et al. (2009) that evaluated the effect of virtual reality intervention on patients' anxiety levels in the preoperative period. An effect size of d=0.920 was obtained by comparing the pre- and post-interventional VAS-A score changes of the intervention group (2.2±2.94) and the control group (5.27±3.69). The G-Power software (G-Power 3.1.9.7, Kiel, Germany) was used for the sample size calculation, applying an effect size of d=0.920, an alpha error probability of 0.05, and a statistical power of (1-β err prob) = 0.95. As a result, a total of 96 patients were enrolled in the study, with 32 patients allocated to each group.

Patients aged ≥ 18 years, scheduled for elective abdominal surgery (including appendectomy, ileal/bowel surgery, hernia repair surgery, gallbladder/pancreas surgery) waiting at the service to be transferred to the operating room in the morning of surgery, and able to communicate and provide informed consent. Patients scheduled to undergo abdominal cancer surgery, those requiring unplanned surgery such as emergency cases, those in isolation, those with visual and/or auditory disabilities, and those with neurological problems such as vertigo were excluded.

In this study, data were collected using "Patient Information Form", "Visual Analog Scale-Anxiety (VAS-A)", and "Smart Bracelet".

ELIGIBILITY:
Inclusion Criteria Patients aged ≥ 18 years

Scheduled for elective abdominal surgery (e.g., appendectomy, ileal/bowel surgery, hernia repair, gallbladder/pancreas surgery)

Awaiting transfer to the operating room on the morning of surgery

Able to communicate effectively

Able to provide informed consent

Exclusion Criteria Patients scheduled for abdominal cancer surgery

Patients undergoing unplanned or emergency surgery

Patients in isolation

Patients with visual and/or auditory impairments

Patients with neurological conditions such as vertigo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Preoperative Anxiety Level-1 | 2 minutes before the intervention. Preoperative.
  Visual Analogue Scale-Anxiety (VAS-A):This scale was used to evaluate patients' preoperative anxiety levels on the morning. It consists of a horizontal line on the paper with scored from "0" for "experiencing no anxiety" on the left side to "10" for " experiencing too much anxiety" on the right side.It is also reported to be valid in evaluating preoperative anxiety of surgery patients. The anxiety levels of a total of 96 patients were evaluated subjectively using the VAS-A scale. Patients marked the level of anxiety they felt on a scale
Preoperative Stress Level-1 | 2 minutes before the intervention. Preoperative.
  This wearable device (smart bracelet) was used to evaluate the stress levels and heart rates of patients. It utilizes a built-in sensor to estimate users' stress levels, providing a score ranging from 1 to 100, where 1 indicates minimal stress and 100 represents very high stress. This estimation is derived from Heart Rate Variability (HRV) data. The device applies a proprietary algorithm-referred to as a stress model-to interpret HRV fluctuations and classify the user's stress level accordingly. The stress levels of a total of 96 patients were measured objectively with a smart bracelet.
Preoperative Heart Rate | 2 minutes before the intervention. Preoperative.
  This wearable device was used to evaluate the stress levels and heart rates of patients. It utilizes a built-in sensor to estimate users' stress levels, providing a score ranging from 1 to 100, where 1 indicates minimal stress and 100 represents very high stress. This estimation is derived from Heart Rate Variability (HRV) data. The device applies a proprietary algorithm-referred to as a stress model-to interpret HRV fluctuations and classify the user's stress level accordingly. The heart rate levels of a total of 96 patients were measured objectively with a smart bracelet.

SECONDARY OUTCOMES:
Preoperative Anxiety Level-2 | Preoperative. immediately after intervention.
  Visual Analogue Scale-Anxiety (VAS-A):This scale was used to evaluate patients' preoperative anxiety levels on the morning. It consists of a horizontal line on the paper with scored from "0" for "experiencing no anxiety" on the left side to "10" for " experiencing too much anxiety" on the right side.It is also reported to be valid in evaluating preoperative anxiety of surgery patients. The anxiety levels of a total of 96 patients were evaluated subjectively using the VAS-A scale. Patients marked the level of anxiety they felt on a scale. The patient was evaluated after watching the video. The average video duration was 20 minutes.
Preoperative Stress Level | Preoperative. immediately after intervention.
  This wearable device was used to evaluate the stress levels and heart rates of patients. It utilizes a built-in sensor to estimate users' stress levels, providing a score ranging from 1 to 100, where 1 indicates minimal stress and 100 represents very high stress. This estimation is derived from Heart Rate Variability (HRV) data. The device applies a proprietary algorithm-referred to as a stress model-to interpret HRV fluctuations and classify the user's stress level accordingly. The patient was evaluated after watching the video. The average video duration was 20 minutes. The stress levels of a total of 96 patients were measured objectively with a smart bracelet.
Preoperative Heart Rate | Preoperative. immediately after intervention.
  This wearable device was used to evaluate the stress levels and heart rates of patients. It utilizes a built-in sensor to estimate users' stress levels, providing a score ranging from 1 to 100, where 1 indicates minimal stress and 100 represents very high stress. This estimation is derived from Heart Rate Variability (HRV) data. The device applies a proprietary algorithm-referred to as a stress model-to interpret HRV fluctuations and classify the user's stress level accordingly. The patient was evaluated after watching the video. The average video duration was 20 minutes. The heart rate levels of a total of 96 patients were measured objectively with a smart bracelet.

CONTACTS AND LOCATIONS:
Overall Officials: Dogan Albayrak, Dr, Principal Investigator — Trakya University
Locations (1):
- Trakya University Hospital, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared when requested from the authors.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: The primary author is reached via e-mail and if requested, data will be shared with the consent of all authors.

REFERENCES:
- [Background] Herrera-Espineira C, Rodriguez del Aguila Mdel M, Rodriguez del Castillo M, Valdivia AF, Sanchez IR. Relationship between anxiety level of patients and their satisfaction with different aspects of healthcare. Health Policy. 2009 Jan;89(1):37-45. doi: 10.1016/j.healthpol.2008.04.012. Epub 2008 Jun 11. PMID 18550203
- [Background] Jlala HA, French JL, Foxall GL, Hardman JG, Bedforth NM. Effect of preoperative multimedia information on perioperative anxiety in patients undergoing procedures under regional anaesthesia. Br J Anaesth. 2010 Mar;104(3):369-74. doi: 10.1093/bja/aeq002. Epub 2010 Feb 1. PMID 20124283
- [Background] Lin LY, Wang RH. Abdominal surgery, pain and anxiety: preoperative nursing intervention. J Adv Nurs. 2005 Aug;51(3):252-60. doi: 10.1111/j.1365-2648.2005.03502.x. PMID 16033593
- [Background] Hendricks TM, Gutierrez CN, Stulak JM, Dearani JA, Miller JD. The Use of Virtual Reality to Reduce Preoperative Anxiety in First-Time Sternotomy Patients: A Randomized Controlled Pilot Trial. Mayo Clin Proc. 2020 Jun;95(6):1148-1157. doi: 10.1016/j.mayocp.2020.02.032. PMID 32498771
- [Background] Mosso JL, Gorini A, De La Cerda G, Obrador T, Almazan A, Mosso D, Nieto JJ, Riva G. Virtual reality on mobile phones to reduce anxiety in outpatient surgery. Stud Health Technol Inform. 2009;142:195-200. PMID 19377147
- See also: video that participants will watch with mobile virtual glasses - also video that participants will watch without virtual glasses — https://www.youtube.com/watch?v=uEMmpJgaXvo&ab_channel=4KRelaxationChannel

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT05718661/Prot_SAP_000.pdf